CLINICAL TRIAL: NCT04158557
Title: Strategies for Management of Knee Osteoarthritis : Innovation and Medico-economic Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: INSERM
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoarthritis is an evolving joint disease caused by degeneration of bones and cartilage, with significant personal and social impact. Osteoarthritis of the knee is the most common type of osteoarthritis, affecting up to 19% of adults (aged 45 and over) according to recent studies.

The costs associated with the management of osteoarthritis involve not only direct treatment strategies (clinical evaluations, drugs, prostheses, surgery), but also significant indirect costs (loss of productivity) The severity of knee osteoarthriris symptoms and the types of interventions are highly variable. There are surgical and nonsurgical treatment strategies. The replacement of the knee joint by a total prosthesis is a surgical choice for severe knee osteoarthritis which currently represents the basic treatment. However, a large proportion of patients with knee osteoarthritis can not or do not wish to have surgery, either because of the unavailability of the choice of surgery, or the disability and post-operative pain that can be caused by surgery.

Since surgery is not always the preferred or available treatment for people with knee osteoarthritis, it has been shown that acting on modifiable risk factors (severe obesity) can significantly reduce the pain and disability but it is not always sufficient.

Other effective therapeutic osteoarthritis strategies include biomechanical interventions, intra-articular injections like corticosteroids ; anti-inflammatory and analgesic drugs, exercise, patient education and bodybuilding. There is also an innovative strategy that is under development and consists of the use of nanostructured and functionalized implants for bone and cartilage regeneration.

The objective of this study is to carry out a medico-economic study centered on knee osteoarthritis management strategies. At a time when the decisions of management of pathologies must be based on the efficiency of the possible therapies, and given the high prevalence of knee osteoarthritis, it appears crucial to carry out this type of study in order to 'bring elements to public health decision makers. In addition, there is a demand for medico-economic assessment of osteoarthritis management strategies emerging in the literature. To carry out this study, we plan to carry out an extensive review of the literature on relevant non-surgical strategies for patients with moderate and severe knee osteoarthritis and for whom total knee replacement was feasible. This will aim to extract data to develop a modeling (Markov models) of knee osteoarthritis management by different therapeutic strategies. At this stage, the cost and quality of life data for the models will be searched in order to be linked to the strategy cost within a medico-economic evaluation.

If the literature proves to be insufficient, the use of the data of the University Hospitals of Strasbourg (retrospective study), the realization of an epidemiological study (prospective study) will be a possible in order to make the model.

ELIGIBILITY:
Inclusion Criteria:

* moderate or severe knee osteoarthritis

Exclusion Criteria:

* another disease than knee osteoarthritis

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: male of female aged from 18 to 85 years with moderate to severe knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline and 12 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is to assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis (OA).
  The WOMAC consists of 24 items divided into 3 subscales:
  * Pain (5 items):
  * Stiffness (2 items):
  * Physical Function (17 items)
  Each scale uses the following descriptors for all items: none, mild moderate, severe, and extreme. These correspond to an ordinal scale of 0-4.
  The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68.
  A total WOMAC score is created by summing the items for all three subscales. (0-96) Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
The Short Form (36) Health Survey (SF-36) | baseline and 12 months
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health

CONTACTS AND LOCATIONS:
Locations (1):
- Inserm-Unistra, Umr 1260, Strasbourg, Alsace, France